CLINICAL TRIAL: NCT06427980
Title: Efficacy and Safety of Chinese Herbal HuoXue LiShui Formula for Chronic Subdural Hematoma: a a Prospective, Randomized, Double-blinded, Placebo-controlled, Multicenter Trail
Brief Title: Efficacy and Safety of Chinese Herbal HuoXue LiShui Formula for Chronic Subdural Hematoma
Acronym: CHARM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Weiming Liu, Professor, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KY2023-265
Record Dates: First submitted 2024-05-20; First posted 2024-05-24 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Chronic Subdural Hematoma
Keywords: Chronic Subdural Hematoma; Chinese herbal formula; HuoXue LiShui; Pharmacotherapy; Randomized controlled trial
MeSH Terms: conditions — Hematoma, Subdural, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The investigators in charge of the recruitment and follow-up evaluation and participants will be blinded, along with the outcome assessors and data analysts.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HXLS group (Experimental): The HXLS granules are produced from four Chinese herbal pieces: Yi Mu Cao (Leonurus heterophyllus, 15.0g), Zhi Shui Zhi (Hirudo, 1.5g), Tao Ren (Semen persicae, 6.0g), and Hong Hua (Carthamus tinctorius L, 6.0g).
  Interventions: Drug: Chinese Herbal formula HuoXue LiShui
- placebo group (Placebo Comparator): The placebo will be consistent with the HXLS oral granules in appearance, taste, and weight, to the greatest extent possible. It included Hu Jing (28.0g)
  Interventions: Drug: Chinese Herbal formula Placebo

INTERVENTIONS:
Drug: Chinese Herbal formula HuoXue LiShui — The intervention consists of the oral administration of granule with either HXLS or a placebo substance, one bag (28.5 g) twice daily after meals for a period of 8 weeks. The granules are produced from four Chinese herbal pieces: Yi Mu Cao (Leonuri Herbal, 15.0g), Zhi Shui Zhi (Hirudo, 1.5g), Tao Ren (Semen persicae, 6.0g), and Hong Hua (Carthami Flos, 6.0g).
  Other Names: HuoXue LiShui
  Arms: HXLS group
Drug: Chinese Herbal formula Placebo — The placebo will be consistent with the HXLS oral granules in appearance, taste, and weight, to the greatest extent possible. In terms of outer packing, the HXLS and placebo granules will be exactly the same. It included Hu Jing (28.5g)
  Other Names: Placebo
  Arms: placebo group

SUMMARY:
A prospective, randomised, double-blind, placebo-controlled, multicentre trial was designed to compare the the incidence of hematoma progression requiring operation or hematoma recurrence requiring re-operation and improves clinical outcomes at 24 weeks in patients with CSDH of treatment in the HXLS and placebo groups.

DETAILED DESCRIPTION:
The CHARM trial is a prospective, randomized, double-blinded, placebo-controlled, multicenter clinical study. The trial aims to investigate the efficacy of the Chinese herbal formula HXLS as an addition to a primary conservative treatment of CSDH in an effort to prevent surgery. The investigators hypothesize that, compared with placebo, the Chinese herbal formula HXLS reduce incidence of hematoma progression requiring operation or hematoma recurrence requiring re-operation and improves clinical outcomes at 24 weeks in patients with CSDH. Consequently, the defined null hypothesis will be that there is no difference between the groups. In total, 160 patients will be randomly assigned to the HXLS group and the placebo group at a 1:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 90 years and either gender will be included.
2. Supratentorial, unilateral or bilateral CSDHs will be verified via cranial CT or magnetic resonance imaging (MRI).
3. Primary hematoma or residual hematoma after burr-hole drainage.
4. Stable vital signs and neurological deficits are indicated by a Glassgow Coma Scale (GCS) score ≥ 14 and a modified Rankin scale (mRS) score ≤ 2.
5. No risk of brain herniation or recent immediate need for surgery will be evaluated by 2 attending neurosurgeons.
6. Written informed consent will be obtained from patients or their next of kins according to their cognitive status.

Exclusion Criteria:

1. Unstable vital signs or symptoms of brain herniation, including severe headache, nausea and vomiting, or disturbed consciousness.
2. Progressive or apparent neurological deficit with a GCS score < 14 or mRS score > 2.
3. Midline shift > 10 mm on the radiological image.
4. Previous medication treatment for CSDH.
5. Previous intracranial surgery for any other neurological disorder.
6. Structural causes for secondary CSDH, including arachnoid cysts, intracranial tumors, vascular malformations, spontaneous intracranial hypotension, coagulopathy, and conversion from acute subdural hematoma.
7. Known hypersensitivity or allergy to HXLS or to any of the ingredients.
8. Malignant tumors.
9. Life expectancy of < 1 year.
10. Abnormal liver function or liver diseases, including uncontrolled hepatitis (alanine transaminase > 120 U/L).
11. Severe renal impairment (estimated glomerular filtration rate < 30 ml/min or serum creatinine > 150 μmol/L).
12. Moderate or severe anemia (hemoglobin ≤ 90 g/L).
13. Severe coagulopathy or a high risk of life-threatening bleeding.
14. Poor medication conditions or the presence of severe comorbidities such that treatment cannot be tolerated or follow-up cannot be completed.
15. Routine oral antithrombotic or antifibrinolytic drugs, steroids, statins, angiotensin-converting enzyme inhibitors, or other traditional Chinese medicines before randomization or are expected to take such medications in the next 24 weeks.
16. Difficulty swallowing oral medication.
17. Pregnancy or lactation.
18. Participating in another study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-03-28 (Estimated)

PRIMARY OUTCOMES:
Rate of operation | From baseline up to 24 weeks after the start of treatment with the study medication
  Surgical rate of hematoma recurrence due to progression of primary hematoma or after burr hole drainage

SECONDARY OUTCOMES:
Chronic subdural hematoma volume | At baseline, and at 4, 8 and 24 weeks
  CSDH volume measured on head CT
Change of Modified Rankin Scale (MRS) between group | At baseline, and at 4, 8, and 24 weeks
  Modified Rankin Scale ranges from score 1 to 6, and higher scores mean a worse clinical outcome, where score 1 indicates normal daily functionality and score 6 indicates death.
Change of Markwalder Grading Scale (MGS) between groups | At baseline, and at 4, 8, and 24 weeks
  Markwalder Grading Scale ranges from grade 0 to 4, and higher scores mean a worse neurological outcome, where grade 0 indicates normal neurological function and grade 4 indicates coma.
Change of Quality of life | At baseline, and at 4, 8, and 24 weeks
  A standardized instrument, EuroQoL 5-Dimension 5-Level (EQ-5D-5L) questionnaire, will be used as a generic measure of health related quality of life. The questionnaire contains 5 dimensions: Mobility, Self-Care, Usual Activities, Pain/Discomfort, and Anxiety/Depression. Each dimension rates across five levels, including 'No problems-Slight problems-Moderate problems-Severe problems-Unable to'.
Change of performance in activities of daily living | At baseline, and at 4, 8, and 24 weeks
  The Barthel Index is scored from 0 to 100. >60 is good, with mild dysfunction, able to perform some activities of daily living independently, and needing some help; 60-41 is moderate. 60-41 is classified as moderate, with moderate dysfunction, requiring a great deal of help to complete activities of daily living; ≤40 is classified as poor, with severe dysfunction, unable to complete most of the activities of daily living or needing help from others.
Change of cognitive functioning | At baseline, and at 4, 8, and 24 weeks
  The Montreal Cognitive Assessment (MOCA) score is an assessment tool designed to facilitate rapid screening for abnormalities in cognitive functioning. It encompasses 11 screening items across eight cognitive domains, including attention and concentration, executive function, memory, language, visual structural skills, abstract thinking, calculation, and orientation. A total score of 30 or above 26 is indicative of normal cognitive function.
Number of falling incidents | At 24 weeks
  Number of falling incidents
Mortality | At 24 weeks
  Mortality
Rate of complications and adverse events between groups | Within 24 weeks
  Rate of complications and adverse events between groups

CONTACTS AND LOCATIONS:
Overall Officials: Weiming Liu, M.D., Principal Investigator — Beijing Tiantan Hospital
Locations (3):
- China (3):
  - Beijing Luhe Hospital, Capital Medical University, Beijing, Beijing Municipality
  - First People's Hospital of Lianyungang, Lianyungang, Jiangsu
  - Beijing Tiantan Hospital, Capital Medical University, Beijing